CLINICAL TRIAL: NCT02652299
Title: Fibrocytes in Early and Longstanding Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Søren Andreas Just, MD, Odense University Hospital
Other Study IDs: S-20140062
Record Dates: First submitted 2015-11-15; First posted 2016-01-11 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Fibrocytes; Synovial biopsy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood, Synovial tissue biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Early Rheumatoid Arthritis group: Following informed written consent, 20 patients with early RA will be enrolled from Odense University Hospital (OUH) during a 12 month period
  Interventions: Biological: Synovial biopsy
- Longstanding Rheumatoid Arthritis group: Following informed written consent, 20 patients with longstanding RA will be enrolled from Odense University Hospital (OUH) during a 12 month period
  Interventions: Biological: Synovial biopsy
- Control group: Synovial tissue and peripheral blood: 20 Non-RA patients who are referred to arthroscopy in a joint of the hand at OUH Department of Orthopedics, Section of hand surgery, are asked to participate by the surgeon at the first ambulatory consultation. Following informed written consent, MRI of hand, a blood sample and synovial biopsies, will be used as control for synovial and plasma fibrocyte levels. The synovial biopsies will be obtained during the planned arthroscopy.
  Interventions: Biological: Synovial biopsy

INTERVENTIONS:
Biological: Synovial biopsy — Synovial tissue for analysis and biobank.

SUMMARY:
This study will focus on a rare cell population called fibrocytes in peripheral blood and synovial tissue in Rheumatoid Arthritis (RA). One group of patients with early RA and one group with long-standing RA. Both groups will be followed for 6 months.

After informed and written consent a control groups is also formed: One for synovial biopsies for patients undergoing a routine arthroscopy, where a peripheral blood sample is also taken.

The hypothesis is that fibrocytes are present in the blood and synovial tissue in RA. Patients with early and long-standing RA have higher concentrations of fibrocytes in peripheral blood and synovial tissue compared to a control groups. Levels of fibrocytes in peripheral blood and synovial tissue are correlated with RA disease activity measures and imaging findings.

DETAILED DESCRIPTION:
The intimal lining of a synovial joint consists of unique cells called fibroblast-like synoviocytes (FLS cells) with interspersed macrophage-like synoviocytes. In the healthy joint macrophage-like synoviocytes are implicated in the innate immune defence and support adaptive immunity, while FLS cells function to regulate the release of nutrients and molecules, including hyaluronan, into the joint cavity.

Rheumatoid arthritis (RA) is a chronic systemic disease with autoimmune traits, which primarily affects synovial joints. The intimal lining of the synovium expands and exhibits characteristics of unregulated growth and loss of contact inhibition. The expanding synovium degrades cartilage and erodes into the bone at the cartilage-bone interface, creating the hallmark of RA, the joint erosion.

The RA FLS cell, has a markedly different phenotype than the healthy cell, and plays a key role in the destructive process by the release of pro-inflammatory cytokines and matrix destructive enzymes. FLS cells expand during the joint destructive process, however, there is minimal mitotic activity. The origin of the expanding FLS population is therefore uncertain.

Possible explanations to this phenomenon could be decreased senescence, migration of mesenchymal stem cells from the circulation, epithelial to mesenchymal cell-transition or expansion of a stem cell pool in the synovium. FLS precursors could also migrate to the synovium through pores in cortical bone, as has been demonstrated in mice with collagen-induced arthritis. In a murine model, it has further been shown that RA FLS cells can spread via the systemic circulation from one joint and attack previously unaffected joints.

A possible FLS cell precursor has been identified in peripheral blood and called fibrocytes. Fibrocytes are spindle-shaped cells that express surface receptors of both stromal and hematopoietic cells. The fibrocytes are a rare (~0.5% of leukocytes) population of bone marrow derived mesenchymal progenitor cells. A combination of markers that distinguish fibrocytes from monocytes, macrophages and fibroblasts has been described. In vitro circulating human peripheral blood mononuclear cells and monocytes (CD14+) can differentiate into fibrocytes. Fibrocytes can differentiate in vitro along multiple mesenchymal lineages into adipocytes, chondrocytes, myofibroblasts and osteoblasts. It is unknown which differentiation pathway occurs in vivo or if multiple differentiation profiles can occur .

Increased numbers of circulating fibrocytes have been found in murine RA models. In a small sample of RA patients (six patients, ten controls), peripheral blood fibrocytes had elevated phosphorylation activation compared to controls, and cells were demonstrated in the synovium. Here fibrocyte activation was correlated with arthritis disease activity (DAS28). In a murine model, activated circulating fibrocytes where found to migrate to arthritis joints in the preclinical phase of the disease, and to accumulate in the FLS cell layer of the synovium. Adoptive transfer of circulating fibrocytes in this murine model, led to worsening of joint disease indicating that circulating fibrocytes are involved in RA joint pathology, possibly as a FLS-cell precursor. Further, fibrocytes have also been implicated in extra articular manifestations of RA, e.g. pericarditis (murine model), atherosclerosis, and interstitial lung disease.

Studies on synovial biopsies have been critical in the understanding of RA pathogenesis. A new method of collecting synovial tissue, ultrasound-guided synovial biopsy is safe and well tolerated by patients and reliable for collecting high quality synovial tissue from large and small joints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed RA (according to 2010 classification criteria) who have been diagnosed ≤ 6 months, and who have at least one swollen joint in hands/fingers.
2. Patients with longstanding RA (>5 years duration).
3. Ability and willingness to give written informed consent and to meet the requirements of this protocol.

Exclusion criteria

1. Age < 18 years.
2. Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis or primary vasculitis.
3. History of or current inflammatory joint disease other than RA (e.g. gout, reactive arthritis, psoriatic arthritis, spondyloarthropathy, Lyme disease).
4. Allergy to local aesthetics.
5. Hereditary or acquired (e.g. Anticoagulant Treatment, apart from low dose aspirin) coagulation abnormality.
6. Prednisolone above 7.5 mg/day
7. Skin pathology at site of joint biopsy.
8. Obesity, BMI > 30.
9. Functional class IV as defined by the criteria for classification of functional status in RA.
10. Heart failure (NYHA class III/IV), immunodeficiency, current or past malignant disease (except for non-melanoma skin cancer), recurrent or chronic infections (viral, fungal or bacterial), inflammatory bowel disease, myeloproliferative disorder or other bone marrow disease.
11. Severe nervous system, liver, pulmonary, renal or endocrine disease (including Type 1 diabetes, stable type 2 diabetes is allowable).
12. Major surgery within 8 weeks. Laboratory exclusion Criteria Platelet count <100 x 109 /L or Haemoglobin <5 mmol/L or White blood cells <3 x 109/L or estimated Glomerular Filtration Rate (eGFR) <60.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following informed written consent, RA patients will be enrolled from Odense University Hospital (OUH) during a 12 month period.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Fibrocytes in the peripheral blood. | 6 months
  Compare level of fibrocytes (Fibrocytes/uL) in peripheral blood between the group of healthy controls and patients with early and long-standing RA.
  Compare level of fibrocytes (Fibrocytes/uL) at start of observation to end of observation in both RA groups.

SECONDARY OUTCOMES:
Interstitial lung disease and fibrocyte level. | 6 months
  Is the fibrocyte level in peripheral blood at presentation correlated with signs of beginning interstitial lung disease, defined as a reduction in the Carbon monoxide diffusion capacity (as mL/min/mm Hg and as a percentage of a predicted value) measured by a lung function test at presentation and at the end of the 6 months period.
Fibrocytes and RA disease activity by imaging, and synovial tissue analysis. | 6 months
  Fibrocyte levels are correlated to disease activity measured by imaging findings on x-ray (Larsen Score), ultrasound (Synovitis and Doppler Score (0-3)) and MRI (RAMRIS score) and degree of synovial that inflammation.

OTHER OUTCOMES:
Fibrocytes in the synovial tissue. | 6 months
  Compare level of fibrocytes in synovial tissue (Fibrocytes/mm3) between healthy controls and RA groups. Compare level of fibrocytes in synovial tissue between RA groups, at start of observation to biopsy at end of observation (time 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Søren Andreas Just, MD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Just SA, Nielsen C, Werlinrud JC, Larsen PV, Hejbol EK, Tenstad HB, Daa Schroder H, Barington T, Torfing T, Humby F, Lindegaard H. Fibrocytes in early and long-standing rheumatoid arthritis: a 6-month trial with repeated synovial biopsy, imaging and lung function test. RMD Open. 2021 Mar;7(1):e001494. doi: 10.1136/rmdopen-2020-001494. PMID 33674419